CLINICAL TRIAL: NCT04576949
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Phase 3 Trial Evaluating the Efficacy and Safety of Cytisinicline in Adult Smokers
Brief Title: A Study of Cytisinicline for Smoking Cessation in Adult Smokers
Acronym: ORCA-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACH-CYT-03
Record Dates: First submitted 2020-09-25; First posted 2020-10-06 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — cytisine; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo + Behavioral Support (Placebo Comparator): one placebo tablet orally (PO) three times daily (TID) plus behavioral support for 12 weeks
  Interventions: Drug: Placebo; Behavioral: Behavioral support
- Cytisinicline + Placebo + Behavioral Support (Experimental): one cytisinicline tablet PO TID plus behavioral support for 6 weeks followed by one placebo tablet PO TID plus behavioral support for 6 weeks
  Interventions: Drug: Cytisinicline; Drug: Placebo; Behavioral: Behavioral support
- Cytisinicline + Behavioral Support (Experimental): one cytisinicline tablet PO TID plus behavioral support for 12 weeks
  Interventions: Drug: Cytisinicline; Behavioral: Behavioral support

INTERVENTIONS:
Drug: Cytisinicline — film-coated oral tablets containing 3 mg cytisinicline
  Other Names: Cytisine
  Arms: Cytisinicline + Behavioral Support; Cytisinicline + Placebo + Behavioral Support
Drug: Placebo — film-coated oral tablets containing matched placebo
  Arms: Cytisinicline + Placebo + Behavioral Support; Placebo + Behavioral Support
Behavioral: Behavioral support — Behavioral support sessions by a qualified study site staff member will be participant-driven and will include direct engagement with the subject about their attempt to quit smoking. Each session will last approximately 10 minutes.

SUMMARY:
This placebo-controlled Phase 3 study is being conducted at sites within the United States to evaluate 3 mg cytisinicline 3 times daily (TID) for treatment duration of 42 days/6 weeks and evaluate 3 mg cytisinicline TID for treatment duration of 84 days/12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age ≥18 years.
2. Current daily cigarette smokers (averaging at least 10 cigarettes per day upon completing a 7-day screening smoking diary) and who intend to quit smoking.
3. Expired air carbon monoxide (CO) ≥10 ppm.
4. Failed at least one previous attempt to stop smoking with or without therapeutic support.
5. Willing to initiate study treatment on the day after randomization and set a quit date within 5-7 days of starting treatment.
6. Willing to actively participate in the study's smoking cessation behavioral support provided throughout the study.
7. Able to fully understand study requirements, willing to participate, and comply with dosing schedule.
8. Sign the Informed Consent Form.

Exclusion Criteria:

1. More than 1 study participant in same household.
2. Previous cytisinicline treatment in a prior clinical study or any other cytisine usage.
3. Known hypersensitivity to cytisinicline or any of the excipients.
4. Positive urinary drugs of abuse screen, determined within 28 days before the first dose of cytisinicline.
5. Clinically significant abnormal serum chemistry or hematology values within 28 days of randomization (ie, requiring treatment or monitoring).
6. Clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined after minimum of 5 minutes in supine position within 28 days of randomization (ie, requiring treatment or further assessment).
7. Body mass index (BMI) classification for being underweight (<18.5 kg/m^2) or having ≥Class 2 obesity (≥35 kg/m^2).
8. Recent history (within 3 months) of acute myocardial infarction, unstable angina, stroke, cerebrovascular incident or hospitalization for congestive heart failure.
9. Current uncontrolled hypertension (blood pressure ≥160/100 mmHg).
10. Documented diagnosis of schizophrenia or bipolar psychiatric illness; currently psychotic.
11. Currently having suicidal ideation or risk for suicide ("Yes" to question 4 or question 5 OR "Yes" to any suicidal behavior question on the Columbia - Suicide Severity Rating Scale [C-SSRS]).
12. Current symptoms of moderate to severe depression (Hospital Anxiety and Depression Scale[HADS] score ≥11).
13. Renal impairment defined as a creatinine clearance (CrCl) <60 mL/min (estimated with the Cockroft-Gault equation).
14. Hepatic impairment defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.0 x the upper limit of normal (ULN).
15. Women who are pregnant or breast-feeding.
16. Male or female subjects of childbearing potential who do not agree to use acceptable methods of birth control during the study treatment period.
17. Participation in a clinical study with an investigational drug in the 4 weeks prior to randomization.
18. Treatment with other smoking cessation medications (bupropion, varenicline, nortriptyline, or any nicotine replacement therapy [NRT]) in the 4 weeks prior to randomization or planned use of these other smoking cessation medications during the study.
19. Use within the 2 weeks prior to randomization or planned use during the study of non-cigarette and/or noncombustible nicotine products (pipe tobacco, cigars, snuff, smokeless tobacco, hookah, e-cigarettes/vaping) or marijuana smoking or vaping.
20. Any other reason that the investigator views the subject should not participate or would be unable to fulfill the requirements for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Rigotti, MD, Principal Investigator — Mass General/Harvard Medical School
Locations (17):
- United States (17):
  - Alliance for Multispecialty Research, LLC., Mobile, Alabama
  - Arizona State University, Phoenix, Arizona
  - Alliance for Multispecialty Research, LLC, Coral Gables, Florida
  - Clinical Research Atlanta, Atlanta, Georgia
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - AMR Lexington, Lexington, Kentucky
  - Alliance for Multispecialty Research, LLC, New Orleans, Louisiana
  - Massachusetts General Hospital - Clinical Genetic Research Facility, Boston, Massachusetts
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - Rochester Clinical Research, Inc., Rochester, New York
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina
  - Alliance for Multispecialty Research, LLC., Knoxville, Tennessee
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Alliance for Multispecialty Research, LLC, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prochaska J, Rubinstein M, Perdok R, Blumenstein B, Jacobs C. Cytisinicline for smoking cessation in individuals with self-reported COPD: a post hoc analysis of the ORCA-2 and ORCA-3 trials. Thorax. 2026 Jan 15;81(2):164-169. doi: 10.1136/thorax-2025-223880. PMID 40962497
- [Derived] Rigotti NA, Benowitz NL, Prochaska J, Leischow S, Nides M, Blumenstein B, Clarke A, Cain D, Jacobs C. Cytisinicline for Smoking Cessation: A Randomized Clinical Trial. JAMA. 2023 Jul 11;330(2):152-160. doi: 10.1001/jama.2023.10042. PMID 37432430

RESULTS

PARTICIPANT FLOW:
Groups:
- 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support: one cytisinicline tablet PO TID plus behavioral support for 6 weeks followed by one placebo tablet PO TID plus behavioral support for 6 weeks
- 12 Week Cytisinicline + Behavioral Support: one cytisinicline tablet PO TID plus behavioral support for 12 weeks
Period: Overall Study
Arm/Group | Placebo + Behavioral Support | 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support | 12 Week Cytisinicline + Behavioral Support
Started (randomized) | 271 | 269 | 270
Completed | 194 | 199 | 225
Not Completed | 77 | 70 | 45
Not completed — Adverse Event | 1 | 3 | 2
Not completed — Withdrawal by Subject | 41 | 26 | 18
Not completed — Physician Decision | 3 | 0 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 29 | 37 | 24
Not completed — Other, Not Specified | 2 | 3 | 1
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Behavioral Support | 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support | 12 Week Cytisinicline + Behavioral Support | Total
Number analyzed (Participants) | 271 | 269 | 270 | 810
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (11.96) | 52.2 (11.15) | 53.3 (11.55) | 52.5 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 148 | 135 | 442
  Male | 112 | 121 | 135 | 368
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 26 | 23 | 68
  Not Hispanic or Latino | 252 | 243 | 247 | 742
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 1 | 4
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 4
  Black or African American | 42 | 40 | 48 | 130
  White | 221 | 222 | 216 | 659
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Smoking Abstinence From Weeks 3 to Week 6
Description: Smoking abstinence as verified by weekly expired carbon monoxide (CO) measurements ≤10 parts per million (ppm).
Time Frame: Weeks 3 to 6
Population: All Randomized Set: all randomized participants. Placebo and 6-week treatment arms only.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Behavioral Support | 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support
Number analyzed (Participants) | 271 | 269
percentage of participants | 4.4 | 25.3
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support; Abstinence from Week 3 to Week 6; Test type: Superiority; p < 0.0001, exact computations — Two-sided, calculated by exact computations with clinical site as a stratifier; Odds Ratio (OR) = 8.00, 95% CI 2-sided [3.94 to 16.25] — Stratified by site
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support; Test type: Superiority; p < 0.0001, Exact computations — Two-sided, derived from marginal odds ratio; Odds Ratio (OR) = 7.30, 95% CI 2-sided [3.92 to 14.38] — Marginal (unadjusted) odds ratio
Statistical Analysis 3: Comparison: Placebo + Behavioral Support vs 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — p-value for difference in proportions; Marginal Difference in Proportions = 0.21, 95% CI 2-sided [0.16 to 0.25]

2. Primary Outcome: Percentage of Participants With Smoking Abstinence From Weeks 9 to Week 12
Description: Smoking abstinence as verified by weekly expired CO measurements ≤10 ppm.
Time Frame: Weeks 9 to 12
Population: All Randomized Set: all randomized participants. Placebo and 12-week treatment arms only.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Behavioral Support | 12 Week Cytisinicline + Behavioral Support
Number analyzed (Participants) | 271 | 270
percentage of participants | 7.0 | 32.6
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs 12 Week Cytisinicline + Behavioral Support; Abstinence from Week 9 to Week 12; Test type: Superiority; p < 0.0001, exact computations — Two-sided, calculated by exact computations with clinical site as a stratifier; Odds Ratio (OR) = 6.29, 95% CI 2-sided [3.69 to 11.57] — Stratified by site
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs 12 Week Cytisinicline + Behavioral Support; Test type: Superiority; p < 0.0001, Exact computations — Two-sided, derived from marginal odds ratio; Odds Ratio (OR) = 6.41, 95% CI 2-sided [3.81 to 11.12] — Marginal (unadjusted) odds ratio
Statistical Analysis 3: Comparison: Placebo + Behavioral Support vs 12 Week Cytisinicline + Behavioral Support; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — p-value for difference in proportions; Marginal Difference in Proportions = 0.26, 95% CI 2-sided [0.20 to 0.30]

3. Secondary Outcome: Percentage of Participants With Continuous Smoking Abstinence From Week 6 to Week 24
Description: Smoking abstinence as verified by expired CO measurements ≤10 ppm. Measurements were weekly from Week 6 to Week 12 and monthly from Week 12 to Week 16.
Time Frame: Week 6 to Week 24
Population: All Randomized Set: all randomized participants. Placebo and 6-week treatment arms only.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Behavioral Support | 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support
Number analyzed (Participants) | 271 | 269
percentage of participants | 2.6 | 8.9
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support; Abstinence from Week 6 to Week 24; Test type: Superiority; p = 0.0016, exact computations — Two-sided, calculated by exact computations with clinical site as a stratifier; Odds Ratio (OR) = 3.67, 95% CI 2-sided [1.50 to 10.24]; Stratified by site
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support; Test type: Superiority; p = 0.0015, Exact computations — Two-sided, derived from marginal odds ratio; Odds Ratio (OR) = 3.69, 95% CI 2-sided [1.61 to 9.36] — Marginal (unadjusted) odds ratio
Statistical Analysis 3: Comparison: Placebo + Behavioral Support vs 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support; Test type: Superiority; p = 0.0015, Cochran-Mantel-Haenszel — p-value for difference in proportions; Marginal Difference in Proportions = 0.06, 95% CI 2-sided [0.03 to 0.09]

4. Secondary Outcome: Percentage of Participants With Continuous Smoking Abstinence From Week 12 to Week 24
Description: Smoking abstinence as verified by expired CO measurements ≤10 ppm. Measurements were monthly from Week 12 to Week 24.
Time Frame: Week 12 to Week 24
Population: All Randomized Set: all randomized participants. Placebo and 12-week treatment arms only.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Behavioral Support | 12 Week Cytisinicline + Behavioral Support
Number analyzed (Participants) | 271 | 270
percentage of participants | 4.8 | 21.1
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs 12 Week Cytisinicline + Behavioral Support; Abstinence from Week 12 to Week 24; Test type: Superiority; p < 0.0001, exact computations — Two-sided, calculated by exact computations with clinical site as a stratifier; Odds Ratio (OR) = 5.32, 95% CI 2-sided [2.81 to 11.09] — Stratified by site
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs 12 Week Cytisinicline + Behavioral Support; Test type: Superiority; p < 0.0001, Exact computations — Two-sided, derived from marginal odds ratio; Odds Ratio (OR) = 5.31, 95% CI 2-sided [2.88 to 10.29] — Marginal (unadjusted) odds ratio
Statistical Analysis 3: Comparison: Placebo + Behavioral Support vs 12 Week Cytisinicline + Behavioral Support; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — p-value for difference in proportions; Marginal Difference in Proportions = 0.16, 95% CI 2-sided [0.11 to 0.20]

5. Secondary Outcome: Percentage of Participants Taking Cytisinicline Who Were Relapse-Free at Week 24
Description: Relapse is defined as participant reported resuming smoking or an expired CO measure ≥ 10ppm. Relapse is defined as a participant having met one of the following: not being abstinent from Weeks 3 to 6; not being abstinent at the Week 12 visit; not abstinent or not self-reported abstinent during the Week 16 to Week 24 follow-up period. (During the follow-up period (Weeks 16 - 24) up to a total of 5 cigarettes could have been smoked.)
Time Frame: Week 24
Population: All Randomized Set: all randomized participants. Participants in the cytisinicline arms.
Measure: Number; unit: percentage of participants
Arm/Group | 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support | 12 Week Cytisinicline + Behavioral Support
Number analyzed (Participants) | 269 | 270
percentage of participants | 10.4 | 13.3
Statistical Analysis 1: Comparison: 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support vs 12 Week Cytisinicline + Behavioral Support; Relapse free from Week 6 to Week 24; Test type: Superiority; p = 0.3484, exact computations — Two-sided, calculated by exact computations with clinical site as a stratifier; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.75 to 2.33] — Stratified by site
Statistical Analysis 2: Comparison: 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support vs 12 Week Cytisinicline + Behavioral Support; Test type: Superiority; p = 0.3514, Exact computations — Two-sided, derived from marginal odds ratio; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.78 to 2.26] — Marginal (unadjusted) odds ratio
Statistical Analysis 3: Comparison: 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support vs 12 Week Cytisinicline + Behavioral Support; Test type: Superiority; p = 0.0317, Zelen's exact test (Pr ≤ P) — p-value for homogeneity across sites

ADVERSE EVENTS:
Time Frame: From randomization (all-cause mortality) or first dose of study drug (adverse events) through Week 24.
Description: Safety Set: all randomized participants who take at least one dose of study drug.
  Treatment emergent adverse events: events that appear during treatment or are present before treatment and subsequently worsen.
Arm/Group | Placebo + Behavioral Support | 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support | 12 Week Cytisinicline + Behavioral Support
All-Cause Mortality (participants affected / at risk) | 0/270 | 1/269 | 0/270
Serious Adverse Events (participants affected / at risk) | 3/270 | 10/269 | 8/270
Other Adverse Events (participants affected / at risk) | 98/270 | 114/269 | 118/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Behavioral Support (N=270) | 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support (N=269) | 12 Week Cytisinicline + Behavioral Support (N=270)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Coronary artery dissection (Cardiac disorders) | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Superior mesenteric artery syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Transient global amnesia (Nervous system disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Behavioral Support (N=270) | 6 Week Cytisinicline + 6 Week Placebo + Behavioral Support (N=269) | 12 Week Cytisinicline + Behavioral Support (N=270)
Constipation (Gastrointestinal disorders) | 3 | 16 | 13
Diarrhoea (Gastrointestinal disorders) | 15 | 10 | 12
Dry mouth (Gastrointestinal disorders) | 3 | 10 | 6
Nausea (Gastrointestinal disorders) | 20 | 16 | 15
Vomiting (Gastrointestinal disorders) | 3 | 3 | 6
Fatigue (General disorders) | 4 | 9 | 9
COVID-19 (Infections and infestations) | 6 | 6 | 9
Sinusitis (Infections and infestations) | 7 | 4 | 3
Urinary tract infection (Infections and infestations) | 3 | 2 | 8
Weight increased (Investigations) | 3 | 6 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 8
Dizziness (Nervous system disorders) | 5 | 12 | 6
Headache (Nervous system disorders) | 22 | 18 | 21
Abnormal dreams (Psychiatric disorders) | 8 | 22 | 21
Anxiety (Psychiatric disorders) | 5 | 7 | 15
Depression (Psychiatric disorders) | 3 | 6 | 3
Insomnia (Psychiatric disorders) | 13 | 23 | 26
Irritability (Psychiatric disorders) | 5 | 8 | 8
Sleep disorder (Psychiatric disorders) | 3 | 6 | 4
Hypertension (Vascular disorders) | 4 | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are bound by requirements outlined in their individual clinical trial agreements with regard to publication of trial results.

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT04576949/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT04576949/SAP_001.pdf